CLINICAL TRIAL: NCT01118520
Title: An Evaluation of the Effect of an Angiotensin-converting Enzyme (ACE) Inhibitor on the Growth Rate of Small Abdominal Aortic Aneurysms.
Brief Title: AARDVARK (Aortic Aneurysmal Regression of Dilation: Value of ACE-Inhibition on RisK)
Acronym: AARDVARK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO1644; 2010-020226-17 (EudraCT Number); 08/109/02 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal aortic aneurysm; ACE Inhibition
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Viacoram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- perindopril (Active Comparator): ACE inhibitor blood pressure lowering agent
  Interventions: Drug: perindopril arginine
- amlodipine (Active Comparator): calcium channel blocker blood pressure lowering agent
  Interventions: Drug: amlodipine 5mgs
- placebo (Placebo Comparator): inactive substance identical in appearance to the othe two comparators
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: perindopril arginine — 10mgs orally daily for the duration of the trial
  Other Names: coversyl arginine
  Arms: perindopril
Drug: amlodipine 5mgs — 5 mgs taken orally daily for the duration of the trial
  Arms: amlodipine
Drug: placebo — one daily
  Arms: placebo

SUMMARY:
Abdominal aortic aneurysms (AAA) are balloon-like swellings of the body's main blood vessel (aorta) as it courses through the abdomen. As a result of the National Aneurysm Screening programme many more of these will be detected. Small AAAs grow slowly and remain a benign condition until the diameter exceeds 2-3 times the diameter of the normal aorta (about 5.5cm in size), when operative repair of the aneurysm is recommended avoiding the potentially fatal event of bursting and bleeding (aneurysm rupture). It is therefore important to identify a strategy to prevent aneurysm growth.

There is a suggestion that the use of a specific drug class, angiotensin converting enzyme (ACE) inhibitors, may reduce the risk of rupture of the larger aneurysms. This trial will assess whether an ACE inhibitor (perindopril) has aneurysm-related benefits, in patients with small AAAs at screening centres in the London area.

The effects of perindopril versus a placebo(dummy) on AAA growth rates will be compared. In addition by comparing the effects of perindopril with the effects of equivalent blood pressure lowering with another non-ACE inhibitor class of drug (amlodipine) on aneurysm growth rate, we can see whether any benefits of perindopril are simply the result of lowering blood pressure. 225 Patients will be assigned to one of these 3 treatments by chance (randomisation).In addition to analysis of the effect of perindopril and blood pressure lowering,the effect of the treatments on quality of life will be assessed. Patients will return at 3-monthly intervals for an ultrasound scan and blood pressure measurements, with questionnaires regarding quality of life at the start and end of the 2-year research period.

An ultrasound scan is a painless test that uses sound waves to create images of organs and structures inside your body.

DETAILED DESCRIPTION:
This trial will investigate the idea that an ACE-inhibitor reduces abdominal aortic aneurysm (AAA) growth rate, in a pilot 3-arm randomised controlled trial (i.e. the study treatment is chosen by random for each patient). The three interventions are ACE-inhibition with perindopril; equivalent blood pressure reduction with amlodipine (a calcium channel blocker) and a placebo tablet. By comparing the effects in the perindopril and amlodipine arms, this design will permit an evaluation of any blood pressure independent effects of perindopril.

Pending results of this pilot trial, we plan to work with the local and National Aneurysm Screening programme to conduct a larger, definitive trial, to investigate the hypothesis that blood pressure reduction with an ACE-inhibitor slows the rate of small AAA growth preferentially compared with other antihypertensive agents.

Secondary research questions in this trial are the effects of perindopril therapy on aneurysm-related death rates, other diseases possibly caused by an AAA and quality of life compared to similar blood pressure lowering effects with amlodipine and placebo.

ELIGIBILITY:
Inclusion criteria:

Willing and able to give written informed consent

Men or women, aged at least 55 years

With AAA 3 to 5.4 cm in diameter by internal or external measurement according to ultrasound

A systolic BP <150mmHg (unless they require and are already receiving an ACE-inhibitor or amlodipine 10mg daily).

Exclusion criteria:

Patients who are already required to take either an ACE-inhibitor or a calcium channel blocker or Angiotensin II blocker (ARB) who cannot be converted to diuretic therapy and/ora 5mg dose of amlodipine for control (ie SBP < 150mmHg) of their BP.

Those with known renal artery stenosis (>50%), or with a serum creatinine of >180µmol/L

Those unable to give informed consent

Those too frail to travel for 3-monthly surveillance will be excluded

Any clinically significant medical condition which, in the opinion of the investigator, may interfere with the study results and or reduce life expectancy to < 2 years

Participation in another trial of an investigational product or device within the previous 30 days

Known allergy or sensitivity to perindopril or amlodipine

Unable or unwilling to comply with the requirements of the study, in the opinion of the investigator.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Powell, MD, Study Director — Imperial College London; Colin Bicknell, FRCS, Study Director — Imperial College London; Deborah Ashby, PhD, Study Director — Imperial College London; Meryl E Davis, FRCS, Principal Investigator — Royal Free Hospital NHS Trust; Mathew Waltham, FRCS, Principal Investigator — Guys Hospital NHS trust; Neil Poulter, FRCP, Study Director — Imperial College London; Christopher Imray, FRCS, Principal Investigator — University Hospitals Coventry & Warwickshire; Dynesh Rittoo, FRCS, Principal Investigator — The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust; Ian Chetter, FRCS, Principal Investigator — Hull University Teaching Hospitals NHS Trust; Sohail Choksy, FRCS, Principal Investigator — East Suffolk and North Essex NHS Foundation Trust; Tim Lees, FRCS, Principal Investigator — The Newcastle Hospitals NHS Foundation Trust; Andrew Thompson, FRCS, Principal Investigator — York Teaching Hospital NHS Foundation Trust; Vince Smyth, FRCS, Principal Investigator — Manchester University NHS Foundation Trust; Shah Nawaz, FRCS, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Andrew Brown, FRCS, Principal Investigator — City Hospitals Sunderland NHS Foundation Trust; Felicity Meyer, FRCS, Principal Investigator — Norfolk and Norwich University Hospitals NHS Foundation Trust
Locations (9):
- United Kingdom (9):
  - The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - Colchester Hospital, Colchester
  - University Hospital Coventry and Warwickshire, Coventry
  - Hull Royal Infirmary, Hull
  - Royal Free Hospital, London
  - St Thomas' Hospital, London
  - St Mary's Hospital, Imperial College Healthcare NHS Trust, London
  - Charing Cross Hospital, Imperial College NHS Trust, London
  - Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Perindopril: 10mgs orally daily for the duration of the trial
- Amlodipine: 5 mgs taken orally daily for the duration of the trial
Period: Overall Study
Arm/Group | Perindopril | Amlodipine | Placebo
Started | 73 | 72 | 79
Completed | 53 | 49 | 59
Not Completed | 20 | 23 | 20
Not completed — AAA repair | 9 | 7 | 9
Not completed — Adverse Event | 3 | 3 | 3
Not completed — Withdrawal by Subject | 8 | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perindopril | Amlodipine | Placebo | Total
Number analyzed (Participants) | 73 | 72 | 79 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (6.9) | 71.5 (6.7) | 70.7 (7.5) | 71.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 5 | 13
  Male | 71 | 66 | 74 | 211
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 73 | 72 | 79 | 224
Number of participants receiving statin treatment [Count of Participants; unit: Participants] | 53 | 45 | 48 | 146
Number of participants with diabetes [Count of Participants; unit: Participants] | 2 | 6 | 8 | 16
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 130.9 (11.5) | 131.9 (13) | 131.7 (12.2) | 131.5 (12.2)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 76.7 (8) | 78.7 (7) | 77.9 (7.6) | 77.7 (7.5)
Abdominal Aortic Aneurysm external longitudinal diameter [Mean (Standard Deviation); unit: cm] | 4.05 (0.65) | 4.03 (0.69) | 4.06 (0.67) | 4.05 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Growth Rate of Abdominal Aortic Aneurysm
Description: Aneurysm growth rate over 2 years, estimated from the sequential AAA diameter measurements (external diameter measured in the longitudinal plane).
Time Frame: Annual rate over the entire period of 24 month
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Perindopril | Amlodipine | Placebo
Number analyzed (Participants) | 73 | 72 | 79
mm | 1.77 (0.02) | 1.81 (0.02) | 1.66 (0.02)
Statistical Analysis 1: Comparison: Perindopril vs Placebo; Test type: Superiority; p = 0.78, Mixed Models Analysis
Statistical Analysis 2: Comparison: Perindopril vs Amlodipine; Test type: Superiority; p = 0.89, Mixed Models Analysis

2. Secondary Outcome: Number of Participants With Aneurysm Related Death
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Perindopril | Amlodipine | Placebo
Number analyzed (Participants) | 73 | 72 | 79
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Perindopril | Amlodipine | Placebo
All-Cause Mortality (participants affected / at risk) | 2/73 | 2/72 | 3/79
Serious Adverse Events (participants affected / at risk) | 19/73 | 12/72 | 16/79
Other Adverse Events (participants affected / at risk) | 7/73 | 8/72 | 9/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perindopril (N=73) | Amlodipine (N=72) | Placebo (N=79)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Angiodisplasia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Rectum biopsy (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal decomperession (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Toe operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Aneurysm embolism (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Prostate transurethal resection (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Bowel resection (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Biopsy penis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Laser prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Appendictomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Lunger cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Adenocarcinoma of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Swelling of legs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture neck of femur (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Angiography (Investigations) | 0 (0) | 1 (1) | 1 (1)
Laryngoscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cytoscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Endoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0)
Angiogram (Investigations) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract surgery (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gallstones (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis of leg (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis of arm (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perindopril (N=73) | Amlodipine (N=72) | Placebo (N=79)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diziness (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Blackout (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Numbness in hands, forearms, elbows (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sweating (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling sick (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling unwell (General disorders) | 1 (1) | 0 (0) | 0 (0)
Upset stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Itchy skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ankle swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Numbness in feet (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Other (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2010-07-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT01118520/Prot_000.pdf